CLINICAL TRIAL: NCT01628471
Title: A Phase I/IIa Dose-Escalation Study of the Decitabine-Genistein Drug Combination in Advanced Solid Tumors and Non-Small Cell Lung Cancer (NSCLC) Subjects
Brief Title: MTD Determination, Safety and Efficacy of the Decitabine-Genistein Drug Combination in Advanced Solid Tumors and Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uman Pharma (Industry)
Collaborators: DSM Nutritional Products, Inc. (Industry); MDEIE Ministry, Québec Government (Unknown); INRS-Institut Armand Frappier , Université du Québec (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMAN-10-01
Record Dates: First submitted 2012-05-09; First posted 2012-06-26 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Phase I b : advanced solid malignancy; Phase II a: stage III b or IV, Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Decitabine; Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine + genistein single arm (Experimental): decitabine injectable, by infusion, 5 ascending doses (60 to 500 mg/m2) genisteine capsules, 3 x 50 mg capsules twice a day
  Interventions: Drug: decitabine in combination with genistein

INTERVENTIONS:
Drug: decitabine in combination with genistein — decitabine IV infusion ( 10 hrs total), doses from 60 to 500 mg/m2 + fixed daily oral dose of 300 mg genisteine

SUMMARY:
Lung cancer is one of the most prevalent and lethal neoplasias in the world. Currently used chemotherapy regimens have been disappointing in improving overall survival. Decitabine is a S-phase pyrimidine analog that induces DNA hypomethylation. This drug is currently used to treat Myelodysplastic Syndrome ( MDS) and has been studied for the treatment of leukemia. Genistein, is a soy extracted non-toxic isoflavone and phytoestrogen, which has been shown to inhibit activity of cell signaling pathways, such as those driven by tyrosine kinases. Results from in vitro experiments unambiguously demonstrated that the combination of these two compounds induces a synergistic reduction of the multiplication of lung, colon, breast and leukemic cancer cells. Consequently, clinical evaluation of this drug combination is warranted in Non Small Cell Lung Cancer ( NSCLC), and it is hypothezised that this new regimen will safely improve overall tumor response rate and cancer progression free survival.

The proposed trial is a two part study: The phase I part is an open-label, dose-escalation evaluation in subjects with advanced solid tumors who have failed standard therapies and for whom no curative therapeutic option exists.

A cohort of three subjects will be treated per dose level. One cycle is 28 days. Five different, increasing dose levels ranging from 60 mg/m2 to 500 mg/m2 of IV decitabine combined with a fixed oral dose of 150 mg BID of genistein will be tested. The Maximum Tolerated Dose (MTD) will be determined based on the occurrence of Dose Limiting Toxicities (DLTs).

In the phase IIa part of the study, only Stage IIIb and IV advanced NSCLC patients will be treated at the recommended decitabine MTD dose combined with genistein. Safety and preliminary efficacy will be assessed. It is expected that a maximum sample of 46 patients will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent.
* Males or females.
* 18-75 years.
* Histologically or cytologically confirmed non-estrogen dependent advanced solid malignancy who has failed standard therapies and/or for which no curative therapeutic option exists (phase I) or ;
* Histologically or cytologically confirmed NSCLC of stage IIIb or IV (phase IIa) that has failed or is ineligible to standard therapies.
* One or more tumor lesions measurable by RECIST criteria
* Life expectancy of at least 3 months.
* ECOG performance of 2 or less.

Exclusion Criteria:

* Prior decitabine or genistein therapy.
* Received cytotoxic agent, hormonal therapy, radiation therapy, or other targeted cancer therapies or investigational agent within 4 weeks prior to study entry.
* Patients with confirmed estrogen receptor-positive cancers, or patients with a primary breast or endometrial cancer for which phenotyping analysis has not been performed.
* Presence of uncontrolled brain metastases or leptomeningeal disease.
* Uncontrolled cardiovascular disorders, including symptomatic heart failure, unstable angina and cardiac arrhythmias.
* Inadequate baseline organ function as shown by following laboratory values :

  * Hemoglobin < 90 g/L
  * Absolute neutrophil count < 1,500 /microliter
  * Platelet count < 100,000 /microliter
  * Total bilirubin > 1.5 ULN
  * AST and ALT > 2.5 ULN
  * Creatinine clearance < 60 ml/min
* To be dependent of oxygen treatment.
* Active infections requiring antibiotics.
* Pregnancy or breastfeeding. All women of child-bearing potential must have a negative pregnancy test prior to first receiving protocol therapy.
* Known allergic reactions to soy derivatives or deoxycytidine derivatives.
* Active alcohol or drug abuse.
* Any co-morbid condition that in the judgment of the investigator renders the subject at high risk of treatment complication or reduces the probability of assessing clinical effect.
* Other malignancies diagnosed within the last 5 years with the exception of Basal Cell Carcinoma of the skin.
* Gastrointestinal disorders or abnormalities that may interfere with the absorption of genistein.
* Patients unable to comply with the study protocol and follow-up schedule for any psychological, familial, sociological or geographical reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 day treatment cycle for MTD assessment; 4-6 cycles to be administered
  MTD determination will based on the incidence of reported adverse events (including dose-limiting toxicities) and abnormal laboratory test results.

SECONDARY OUTCOMES:
To determine the drug plasma concentrations of decitabine and genistein. | Up to 6 , 28 day treatment cycles
  Plasma drug levels will be used to obtain preliminary PK profile. Up to 11 blood samples to be obtained from each enrolled patient, over several cycles.
Preliminary clinical efficacy assessment | Up to 6, 28 day treatment cycles
  Preliminary efficacy of the investigational regimen will include the assessment of Overall Response Rate ( ORR) and Progression Free Survival(PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Normand Blais, MD, FRCP(C), Principal Investigator — Hôpital Notre Dame du CHUM
Locations (1):
- Hôpital Notre Dame du CHUM, Montreal, Quebec, Canada

REFERENCES:
- See also: Study sponsor — http://www.umanpharma.com